CLINICAL TRIAL: NCT01482286
Title: Effect of Weight and Insulin Sensitivity on Reproductive Function in PCOS
Acronym: PULSE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment and enrollment.
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC11016; R00HD060762 (NIH)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Exercise; Diet; Insulin resistance; Weight
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity; Insulin Resistance; Body Weight | interventions — Metformin; Diet Therapy; Caloric Restriction; Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Metformin (Experimental): Subjects randomized to the metformin treatment group will receive 1000 mg extended release metformin hydrochloride tablets (Bristol Myers Squibb) twice per day with food approximately 8 hours apart.
  Interventions: Drug: Metformin
- Dietary Restriction (Experimental): Subjects randomized to the dietary restriction group (DR) will reduce their energy intake by 25% from their weight maintenance energy intake determined at baseline by doubly labeled water.There will be no gradual ramping of dietary restriction. The 25% energy reduction goal will apply from the first day of the intervention for a period of 24 weeks. Subjects will be asked to not modify their normal level of physical activity.
  Interventions: Behavioral: Dietary Restriction
- Exercise (Experimental): Subjects randomized to the exercise training group will complete a structured program of aerobic training 3 to 4 times per week and resistance exercises 2 times per week.
  Interventions: Behavioral: Exercise Training
- Control (No Intervention): Subjects randomized to the no treatment control group will be asked to continue, as normal their usual dietary and exercise regimen. Subjects will be asked to not begin diet or exercise regimens through the 24-week study or to begin medical treatment for PCOS.

INTERVENTIONS:
Drug: Metformin — Subjects randomized to the metformin treatment group will receive 1000 mg extended release metformin hydrochloride tablets (Bristol Myers Squibb) twice per day with food approximately 8 hours apart.
  Other Names: metformin hydrochloride tablets
  Arms: Metformin
Behavioral: Dietary Restriction — Subjects randomized to the dietary restriction group will reduce their energy intake by 25% of their weight maintenance energy intake determined at baseline. Total energy expenditure as measured by a 14-day doubly labeled water (DLW) study will be used to determine the baseline energy intake of each subject. There will be no gradual ramping of dietary restriction. The 25% energy reduction goal will apply from the first day of the intervention for a period of 24 weeks. Subjects will be asked to not modify their normal level of physical activity.
  Other Names: 25% DR; Calorie restriction
  Arms: Dietary Restriction
Behavioral: Exercise Training — For the aerobic training component, subjects are required to meet a weekly energy expenditure target of 10 kcal per kg of body weight per week (KKW).
  The resistance training program will be performed 2 days a week. The resistance program includes 9 exercises. The 9 primary exercises are seated chest press, seated row, shoulder press, lat pull down, double leg press, leg extension, leg curl, back extension and abdominal crunch.
  Other Names: Aerobic and resistance training
  Arms: Exercise

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common reproductive disorder in women of reproductive age and despite decades of research the etiology the disorder is not known. The characteristic hyperandrogenism and anovulation is associated with abnormal neuroendocrine function and insulin resistance. Obesity is a common correlated phenotype of Polycystic ovary syndrome and weight gain worsens the reproductive and metabolic complications. Currently there is no evidence-based treatment plan for infertility in Polycystic ovary syndrome; yet weight loss by dietary restriction and regular exercise are strongly advocated. Weight loss and increased insulin sensitivity appear to drive improvements in reproductive outcomes in women with Polycystic ovary syndrome; however, the mechanism connecting these changes with the reproductive axis is not fully understood.

DETAILED DESCRIPTION:
The goal of this study is to determine (using dietary restriction, exercise training, metformin or no treatment), the effects of weight loss and/or improved insulin sensitivity on reproductive function (neuroendocrine and ovarian) in obese women with Polycystic ovary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 40 years, inclusive
* Body mass index ≥ 25 kg/m2
* History of irregular menstrual cycles (fewer than 6 cycles in the past year)
* Clinical and/or biochemical androgen excess (Free androgen index>3.85 and/or hirsuitism rating ≥8)
* Anovulatory menstrual cycles (determined during screening)

Exclusion Criteria:

* Ovulatory menstrual cycles (determined during screening by luteal phase serum progesterone >3ng/mL)
* History or clinical appearance of cardiovascular disease, diabetes (Type 1 or Type 2) and any other significant reproductive, metabolic, hematologic, pulmonary, gastrointestinal, neurologic, immune, hepatic, renal, urologic disorders, or cancer.
* Hemoglobin, hematocrit, red blood cell count, or iron level below the lower limit of normal at the screening visit confirmed by a test repeated within two weeks
* Regular use of medications for weight control, glucose intolerance, thyroid disease
* Use of hormonal contraception containing medroxyprogesterone acetate (A 3 month washout period will be permitted for oral, vaginal and transdermal contraceptives).

Psychiatric and Behavioral Exclusion Criteria

* Smoking
* History of drug or alcohol abuse (up to 14 drinks a week are allowed) within the past two years
* History or presence of an eating disorder as determined by Interview for Diagnosis of Eating Disorders (IDED-IV)
* Beck Depression Index (BDI) score of ≥15 at screening or baseline

Other Exclusion Criteria

* Individuals who have lost more than 5kg (11lbs) in the past 6 months
* Individuals who are pregnant or breast-feeding or whom become pregnant during the study
* Individuals engaged in a regular program of physical fitness involving some heavy physical activity (e.g., jogging or riding fast on a bicycle for 30 minutes or more) at least five times per week over the past year
* Individuals who have metallic objects in their body
* Individuals who donated blood within 30 days prior to the date of randomization
* Individuals unwilling to be assigned at random to either one of the intervention groups
* Unwilling or unable to adhere to the rigors of the data collection (determined by food and activities diaries at screening, see below) and clinical evaluation schedule over the entire 24 week intervention period
* Individuals who plan to move out of the area within the next 12 months or plan to be out of the study area for more than 4 weeks in the next 12 months
* Individuals who reside too far from Pennington

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Broskey NT, Tam CS, Sutton EF, Altazan AD, Burton JH, Ravussin E, Redman LM. Metabolic inflexibility in women with PCOS is similar to women with type 2 diabetes. Nutr Metab (Lond). 2018 Oct 20;15:75. doi: 10.1186/s12986-018-0312-9. eCollection 2018. PMID 30377436
- [Derived] Broskey NT, Klempel MC, Gilmore LA, Sutton EF, Altazan AD, Burton JH, Ravussin E, Redman LM. Assessing Energy Requirements in Women With Polycystic Ovary Syndrome: A Comparison Against Doubly Labeled Water. J Clin Endocrinol Metab. 2017 Jun 1;102(6):1951-1959. doi: 10.1210/jc.2017-00459. PMID 28323951
- See also: Press Release: New Study at Pennington Biomedical Research Center Designed to Identify Factors Affecting Infertility in Women — http://www.pbrc.edu/news/?ArticleID=134
- See also: Study information and how to participate — http://www.pbrc.edu/clinical-trials/current-studies/?studyid=124

RESULTS

PARTICIPANT FLOW:
Groups:
- Dietary Restriction: Subjects randomized to the dietary restriction group (DR) will reduce their energy intake by 25% from their weight maintenance energy intake determined at baseline by doubly labeled water.There will be no gradual ramping of dietary restriction. The 25% energy reduction goal will apply from the first day of the intervention for a period of 24 weeks. Subjects will be asked to not modify their normal level of physical activity.
  Dietary Restriction: Subjects randomized to the dietary restriction group will reduce their energy intake by 25% of their weight maintenance energy intake determined at baseline. Total energy expenditure as measured by a 14-day doubly labeled water (DLW) study will be used to determine the baseline energy intake of each subject. There will be no gradual ramping of dietary restriction. The 25% energy reduction goal will apply from the first day of the intervention for a period of 24 weeks. Subjects will be asked to not modify their normal level of physical ac
- Exercise: Subjects randomized to the exercise training group will complete a structured program of aerobic training 3 to 4 times per week and resistance exercises 2 times per week.
  Exercise Training: For the aerobic training component, subjects are required to meet a weekly energy expenditure target of 10 kcal per kg of body weight per week (KKW).
  The resistance training program will be performed 2 days a week. The resistance program includes 9 exercises. The 9 primary exercises are seated chest press, seated row, shoulder press, lat pull down, double leg press, leg extension, leg curl, back extension and abdominal crunch.
Period: Overall Study
Arm/Group | Metformin | Dietary Restriction | Exercise | Control
Started | 7 | 7 | 8 | 10
Completed | 4 | 4 | 4 | 5
Not Completed | 3 | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Dietary Restriction | Exercise | Control | Total
Number analyzed (Participants) | 7 | 7 | 8 | 10 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (5.0) | 31.3 (6.2) | 29.1 (3.8) | 27.6 (5.6) | 28.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 10 | 32
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 8 | 9 | 29
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 2 | 6 | 18
  White | 3 | 1 | 6 | 4 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Luteinizing Hormone (LH) Pulse Frequency
Description: Change in Luteinizing Hormone (LH) Pulse Frequency measured over a 12-hour period (7:00 PM - 7:00 AM).
  The Mean and Standard Deviation (SD) are the number of pulses recorded on the 12-hour period (7:00 PM - 7:00 AM) and presented as the change from baseline to week 24.
  Only participants who completed the PULSE trial are included in present outcome measure as the primary outcome was established as change from pre-to-post-intervention LF pulse frequency.
Time Frame: Baseline and Week 24
Population: Study stopped due to poor recruitment, enrollment, and retention.
Measure: Mean (Standard Deviation); unit: Number of pulses
Arm/Group | Metformin | Dietary Restriction | Exercise | Control
Number analyzed (Participants) | 4 | 4 | 4 | 5
Number of pulses | -4.0 (11.3) | -1.5 (7.0) | -6.5 (13.4) | -3.0 (2.6)

2. Secondary Outcome: Insulin Sensitivity Expressed as Glucose Disposal Rate (GDR)
Description: Change in insulin sensitivity measured by the euglycemic hyperinsulinemic clamp.
  Unit of measure established as glucose disposal rate (GDR) adjusted to account for kilograms of fat-free mass (FFM)+17.7 per minute to reflect the amount of exogenous glucose necessary to fully compensate for hyperinsulinemia and expressed as a function of metabolic body size.
  Only participants who completed the PULSE trial are included in present outcome measure as the primary outcome was established as change from pre-to-post-intervention Insulin Sensitivity expressed as Glucose Disposal Rate.
Time Frame: Baseline and Week 24
Population: Study stopped due to poor recruitment, enrollment, and retention.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Metformin | Dietary Restriction | Exercise | Control
Number analyzed (Participants) | 4 | 4 | 4 | 5
mg/kg/min | -1.8 (5.5) | 1.0 (1.7) | 0.8 (0.9) | 22.4 (3.3)

ADVERSE EVENTS:
Arm/Group | Metformin | Dietary Restriction | Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 5/7 | 5/7 | 5/8 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=7) | Dietary Restriction (N=7) | Exercise (N=8) | Control (N=10)
Hospitalized (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=7) | Dietary Restriction (N=7) | Exercise (N=8) | Control (N=10)
Edema (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 2 (2) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Excess Gas
Nausea/Vomiting (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0) | 2 (2)
Nonspecific (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomach Virus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Menstrual Complaints (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Ovarian Disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection/Cystitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vaginal Irritation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Yeast Infection (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Ovarian Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Clot (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arm Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Car Accident
Sciatic Nerve Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck/Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache/Migraine (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever/Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu-Like Symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Non-Specific or Surgical
Nosebleed (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore Throat (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) — Watery Eyes or Clear Nasal Drainage
Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Allergies (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Earache (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nonspecific (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No